CLINICAL TRIAL: NCT03303755
Title: Elaboration, Development and Validation of Predictive Models of Weight and Height for the Evaluation of the Growth of Children and Adolescents With Cerebral Palsy
Brief Title: Predictive Models of Weight and Height for the Evaluation of the Growth of Children and Adolescents With Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: National Council of Scientific and Technical Research, Argentina (Other Government)
Collaborators: Universidad Nacional de Córdoba (Other)
Responsible Party: Principal Investigator, Eduardo Cuestas, PhD Reasercher, National Council of Scientific and Technical Research, Argentina
Other Study IDs: IS001087
Record Dates: First submitted 2017-09-14; First posted 2017-10-06 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Cerebral Palsy; Growth; Child
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cerebral palsy (CP) is the most frequent disability in children. The vast majority of these patients are malnourished. In this population, there are practical difficulties to perform a nutritional and growth assessment which makes it difficult to treat and follow up, because of the lack of reference growth in Argentina, and the difficulty in taking anthropometric measurements of weight and height because of their motor compromise, posture and muscle tone.

The main objective is to design and validate predictive models for the nutritional and growth assessment of children and adolescents with CP and instruments for estimating weight and height from body segments, in order to improve care, quality of life of these patients to promote their social inclusion.

Material and method: It will be an observational, descriptive and cross-sectional study. There will be two parts of the study, in the first part the population will be healthy children from 2 to 18 years old from Cordoba, Argentina. The sample size was calculated based on growth WHO standards data, for α=0.05 and 1-β=0.80, creating an stratified sampling divided in 16 age groups for each age. This first part will help to establish which body segments to use.

In the second part, the population will be children and adolescents from 2 to 18 years old with diagnosis of CP from Córdoba, Argentina. A stratified sequential sampling shall be performed. The sample size will be 192 patients, 12 per age stratum. The variables studied will be: weight, height, body segments, sex, age, CP type, feeding path and type of feeding.

For the analysis of the data the normal continuous variables will be described in means with their respective standard deviations and those of non-normal distribution in medians with their ranges. For the development of the predictive equations using body segments measures, a generalizable linear regression model will be used. The correlation coefficient r, determination R2 and test of F will be calculated with p <0.05. To generate predictive growth models, the percentiles from 3 to 97 will be calculated, using the LMS method and a q-q graph.

DETAILED DESCRIPTION:
The aim is to design predictive models of weight and height, through predictive equations using segmental measurements and to develop specific growth patterns, for the nutritional and growth evaluation of children and adolescents with cerebral palsy from different provinces of Argentina.

This research is a cross-sectional study, which consisted of two stages. First, data were collected from children and adolescents aged 2 to 18 years with typical development from which the anthropometric variables associated with weight and height were determined and then used for the analysis of the population with CP. A stratified sampling was made with 17 strata according to age for each sex, pre-establishing a minimum of 20 children for each stratum. Data were collected transversely in two hospitals and two schools in the City of Córdoba until all strata were completed.

In a second stage, data is collected from children and adolescents diagnosed with CP between the ages of 2 and 19 years. Data were included from 17 rehabilitation centers and therapeutic educational centers in 5 provinces of the country (Córdoba, Buenos Aires (CABA), Jujuy, Santiago del Estero and Catamarca). A sequential non-probabilistic sampling was made, including all possible cases of each participating institution. The variables studied were demographic variables, anthropometric measures, nutritional status, type of malnutrition and in the case of the population with PC also variables such as data on access to health, diagnosis, co-morbidities and feeding were included. Normal continuous variables were described as mean and standard deviations, while those of non-normal distribution in medians with their interquartile ranges. Variables are compared by means of t-test or Mann-Whitney as appropriate. Categorical data are expressed in percentages with a 95% confidence interval [95% CI]. To analyze association between variables, Chi square of Mantel-Haentzel was calculated, and OR with its 95% CI. For the development of predictive equations, a generalizable linear regression model will be used. The correlation coefficient r, determination R2 and F test were calculated with a p <0.05. Growth patterns were made using the Generalized Additive Models for Location Scale and Shape (GAMLSS) method. Nutritional status was assessed using the WHO Anthro Plus V1.0.4 program using the WHO standards (2007). The approval of the local ethics committee was obtained and written informed consent was obtained from the participants.

The study of nutrition in patients with PC is an emerging field, for which this work plan seeks to develop methodologies that promote social inclusion by making substantial and necessary contributions to improve the treatment of this pathology.

ELIGIBILITY:
Inclusion Criteria:

* Children with diagnosis of cerebral palsy

Exclusion Criteria:

* children with endocrine or metabolic disorders, genetic diseases and other congenital anomalies that affect or have affected their growth or nutritional status.

Ages: 2 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The population of this study will be made up of children aged 2 to 18 years with a diagnosis of PCs who attend public and private health institutions in Córdoba.
Sampling Method: Non-Probability Sample
Enrollment: 388 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Weight in children | 2 year
  weight in kilograms
Height in children | 2 year
  height in centimeters

SECONDARY OUTCOMES:
Estimated weight | 1 year
  weight in kilograms using Mid Arm Circumference in centimeters
estimated height | 1 year
  height in centimeters using Knee hell height in centimeters

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Cuestas, PhD MD, Study Director — Instituto de Investigaciones en Ciencias de la Salud
Locations (1):
- Instituto de Investigaciones en Ciencias de la Salud, Argentina, Córdoba, Argentina

IPD SHARING:
Plan to Share IPD: Undecided
the research group is yet not decided to make individual participant data available, we wont to have a bigger data base to decide.

REFERENCES:
- [Background] Abdel-Rahman SM, Ahlers N, Holmes A, Wright K, Harris A, Weigel J, Hill T, Baird K, Michaels M, Kearns GL. Validation of an improved pediatric weight estimation strategy. J Pediatr Pharmacol Ther. 2013 Apr;18(2):112-21. doi: 10.5863/1551-6776-18.2.112. PMID 23798905
- [Background] Brooks J, Day S, Shavelle R, Strauss D. Low weight, morbidity, and mortality in children with cerebral palsy: new clinical growth charts. Pediatrics. 2011 Aug;128(2):e299-307. doi: 10.1542/peds.2010-2801. Epub 2011 Jul 18. PMID 21768315
- [Background] Le Roy O. C, Rebollo G. MJ, Moraga M. F, Díaz Sm. X, Castillo-Durán C. Nutrición del niño con enfermedades neurológicas prevalentes. Rev Chil Pediatr. 2010;81(2):103-113.
- [Background] Day SM, Strauss DJ, Vachon PJ, Rosenbloom L, Shavelle RM, Wu YW. Growth patterns in a population of children and adolescents with cerebral palsy. Dev Med Child Neurol. 2007 Mar;49(3):167-71. doi: 10.1111/j.1469-8749.2007.00167.x. PMID 17355471
- [Background] Vega-Sanchez R, de la Luz Gomez-Aguilar M, Haua K, Rozada G. Weight-based nutritional diagnosis of Mexican children and adolescents with neuromotor disabilities. BMC Res Notes. 2012 Jul 4;5:218. doi: 10.1186/1756-0500-5-218. PMID 22559790
- [Background] Bell KL, Davies PS. Prediction of height from knee height in children with cerebral palsy and non-disabled children. Ann Hum Biol. 2006 Jul-Aug;33(4):493-9. doi: 10.1080/03014460600814028. PMID 17060071
- [Background] Kong CK, Wong HS. Weight-for-height values and limb anthropometric composition of tube-fed children with quadriplegic cerebral palsy. Pediatrics. 2005 Dec;116(6):e839-45. doi: 10.1542/peds.2005-1029. PMID 16322142
- [Background] Neela J, Raman L, Balakrishna N, Rao KV. Usefulness of calf circumference as a measure for screening low birth weight infants. Indian Pediatr. 1991 Aug;28(8):881-4. PMID 1808075
- See also: Rosenbaum P, Paneth N, Leviton A, et al. 2007 Definition of CP. Dev Med Child Neurol Suppl. 2007;109(April):8-14 — http://onlinelibrary.wiley.com/doi/10.1111/j.1469-8749.2007.tb12610.x/pdf